CLINICAL TRIAL: NCT02467673
Title: Nanoparticulate Versus Micronized Steroids Delivery for Transdermal Hormone Replacement Therapy: Effects on Blood Pressure, Insulin and C-reactive Protein and in Postmenopausal Women
Brief Title: Nanoparticulate Versus Micronized Steroids Delivery for Transdermal Hormone Replacement Therapy
Acronym: Nanoparticle
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Potiguar (Other)
Collaborators: InBios International, Inc. (Industry); Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, MARCO BOTELHO, PhD, University Potiguar
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Evidence/Unifesp
Record Dates: First submitted 2015-06-07; First posted 2015-06-10 (Estimated); Last update posted 2016-05-24 (Estimated); Status verified 2016-05

CONDITIONS: Menopausal Syndrome
MeSH Terms: interventions — Progesterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- NANOPARTICULATE estradiol+ progesterone (Active Comparator): The Blood samples are collected from the subjects early in the morning after an overnight fast. After serum testing, the identification hormone deficiencies, was determined and then, if necessary, additional transdermal nanostructured estradiol and progesterone is prescribed.
  The patients are evaluated 3 months after THRT treatment protocol. All the patients were instructed about how to use the pump for transdermal application, the first application is performed in the presence of an experienced physician, in order to guarantee standardization and correct use of the THRT. Compliance was defined as completing seventy percent or more of the transdermal applications.
  Interventions: Drug: Nanoparticulate estradiol + progesterone
- MICRONIZED estradiol+ progesterone (Active Comparator): The Blood samples are collected from the subjects early in the morning after an overnight fast. After serum testing, the identification hormone deficiencies, was determined and then, if necessary, additional transdermal micronized estradiol and progesterone is prescribed.
  The patients are evaluated 3 months after THRT treatment protocol. All the patients were instructed about how to use the pump for transdermal application, the first application is performed in the presence of an experienced physician, in order to guarantee standardization and correct use of the THRT. Compliance was defined as completing seventy percent or more of the transdermal applications.
  Interventions: Drug: Micronized estradiol + progesterone

INTERVENTIONS:
Drug: Micronized estradiol + progesterone — Administration of micronized estradiol + progesterone daily by a metered-dose pump during 12 weeks in postmenopausal women with no clinical evidence of cardiovascular disease.
  Other Names: Mic Group
  Arms: MICRONIZED estradiol+ progesterone
Drug: Nanoparticulate estradiol + progesterone — Administration of nanoparticulate estradiol + progesterone daily by a metered-dose pump during 12 weeks in postmenopausal women with no clinical evidence of cardiovascular disease.
  Other Names: NANO Group
  Arms: NANOPARTICULATE estradiol+ progesterone

SUMMARY:
The study aims to asses the effects of micronized (MIC) and nanoparticulate (NANO) transdermal hormone therapy (THT) on blood pressure, ultra-sensitive C-reactive protein (CRP), and cardiovascular risk factors in postmenopausal women.

DETAILED DESCRIPTION:
In this open label study, 27 postmenopausal women, with no clinical evidence of cardiovascular disease, were randomly divided in two groups.

During 12 weeks,

15 patients received on the left forearm micronized (MIC) THT (micronized 17β-estradiol 2.5 mg/day + progesterone 100 mg/day).

and

14 patients received a nanoparticulate (NANO) THT (nanoparticulate 17β-estradiol 2.5 mg/day + progesterone 100mg/day).

After 12 weeks of treatment patients were evaluated.

Baseline and Post-THT measures were determined: Insulin, body mass index, waist circumference, blood pressure, CRP-stratified levels, total testosterone, TSH and FSH levels.

ELIGIBILITY:
Inclusion Criteria:

* A body mass index between 18 and 27 kg/m2;
* Sex live complaints;
* No evidence of cardiovascular disease;
* General good health based on history and physical examination.

Exclusion Criteria:

* A past history of neurological disorder;
* Had received pharmacotherapy for cardiovascular disease before screening
* Taking medication known to interfere with steroids;
* Recent psychiatric or systemic illness;
* Uncontrolled hypertension (blood pressure>160/95mmHg),
* Unstable cardiovascular disease;
* Genital bleeding;
* Use of psychoactive medications,
* Alcohol excess consumption or any other drug abuse;

Ages: 42 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2012-01; Primary Completion 2012-03 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Blood Pressure variation | 12 weeks

SECONDARY OUTCOMES:
C-reactive protein levels after treatment | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ivaldo Silva, PHD, Study Director — Federal University of São Paulo
Locations (3):
- Brazil (3):
  - Gynelogical Center, Fortaleza, Ceará
  - University Potiguar, Natal, Rio Grande do Norte
  - Marco Botelho, São Paulo, São Paulo

REFERENCES:
- [Background] Botelho MA, Martins JG, Ruela RS, Queiroz DB, Ruela WS. Nanotechnology in ligature-induced periodontitis: protective effect of a doxycycline gel with nanoparticules. J Appl Oral Sci. 2010 Jul-Aug;18(4):335-42. doi: 10.1590/s1678-77572010000400003. PMID 20835566
- [Result] Botelho MA, Queiroz DB, Barros G, Guerreiro S, Fechine P, Umbelino S, Lyra A, Borges B, Freitas A, Queiroz DC, Ruela R, Almeida JG, Quintans L Jr. Nanostructured transdermal hormone replacement therapy for relieving menopausal symptoms: a confocal Raman spectroscopy study. Clinics (Sao Paulo). 2014 Feb;69(2):75-82. doi: 10.6061/clinics/2014(02)01. PMID 24519196